CLINICAL TRIAL: NCT00746200
Title: Randomised Controlled Trial of Acupuncture for Patients With Chronic Constipation
Brief Title: Acupuncture for Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chien-Hsun Huang, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200801047R
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Constipation
Keywords: chronic constipation; electroacupuncture; randomized controlled trial
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Procedure: (electro)acupuncture
- S (Sham Comparator)
  Interventions: Procedure: sham acupuncture

INTERVENTIONS:
Procedure: (electro)acupuncture — Frequency of electrostimulation: 15Hz; Duration of electrostimulation: 20min;
  Other Names: electroacupuncture
  Arms: A
Procedure: sham acupuncture — Superficial acupuncture needle stimulation at non-acupoints with TENS applied for seconds
  Arms: S

SUMMARY:
Since there have been few advances for constipation in laxative treatment in the last 50 years, this study is designed to evaluate the efficacy and safety of acupuncture for patients with chronic constipation based on the theory of traditional Chinese Medicine.

DETAILED DESCRIPTION:
Although many people regard regular defecation as important factor to maintain healthy, constipation is still a common problem in general population. Because the symptoms cause serious impairment of life quality, laxatives are commonly prescribed for people and over prescribing of laxatives is also common. Despite the large sums spent on laxatives, there have been few advances in laxative treatment in the last 50 years and there have been minimal research addressing the problem.

Since there is unsatisfactory effect by current pharmacologic therapies and preventive strategies, we look forward to the practice of traditional Chinese medicine, which had abundant clinical experiences and medical records in the past of thousands years ago. Therefore we aim to do the research to create the evidence of acupuncture on the safety, efficacy and quality of life for chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* men or non-pregnant women who are at least 20 years old
* who meet any one of the following three criteria: 1.the one who meets RomeIII criteria; 2.at least once a week of enema/suppository in past three months; 3.laxative use in more than half time of last three months

Exclusion Criteria:

* known colorectal cancer, anal abscess, anal fissure, rectocele, inflammatory bowel disease, megacolon or mechanical bowel obstruction
* unknown cause of gastrointestinal bleeding or acute infection
* history of alcohol or drug abuser
* women who are pregnant, as determined by a urine pregnancy test
* history of adverse reaction to (electro)acupuncture
* received herb or acupuncture therapy within one month prior to enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
score of questionnaire of constipation symptoms | every month

SECONDARY OUTCOMES:
score of questionnaire of quality of life | every month
amount of laxative use | every week
frequency of enema/suppository use/digital maneuver | every week
stool amount | every week
stool consistency | every week
overall efficacy | 2 month
safety (adverse event) | every week
frequency of spontaneous bowel movement | every week

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsun Huang, MD, MSc, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Yun-Lin Branch, Douliu, Taiwan

REFERENCES:
- [Background] Lembo A, Camilleri M. Chronic constipation. N Engl J Med. 2003 Oct 2;349(14):1360-8. doi: 10.1056/NEJMra020995. No abstract available. PMID 14523145